CLINICAL TRIAL: NCT04854629
Title: Effects of the "Spinomed Active" Orthosis on Chronic Back Pain in Women With Osteoporotic Vertebral Bone Fracture and Hyperkyphosis.
Brief Title: Effects of the "Spinomed Active" Orthosis on Chronic Back Pain in Women With Vertebral Fractures.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: medi GmbH & Co. KG, Bayreuth, Germany (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Orthosis Spinomed active
Record Dates: First submitted 2021-04-13; First posted 2021-04-22 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Osteopenia; Kyphosis
MeSH Terms: conditions — Bone Diseases, Metabolic; Kyphosis

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with two study groups in parallel: (1) Spinomed active orthosis or 16 weeks (2) non spinomed active orthosis control
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor were unaware of participant status (i.e. spinomed active or control) and were not allowed to ask correspondingly
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spinomed active orthosis (Experimental): Wearing the orthosis for 16 weeks
  Interventions: Other: Spinomed active
- Control group (No Intervention): No intervention: non spinomed active control

INTERVENTIONS:
Other: Spinomed active — Wearing of the orthosis 2-3 h/twice a day for 16 weeks Supplementation of a maximum of 1000 mg/d calcium and 800 IE/d vitamin D
  Arms: Spinomed active orthosis

SUMMARY:
Osteoporotic vertebral fractures often lead to postural changes, chronic spinal pain conditions and limited functionality. Orthoses that straighten the spine have been shown in studies to have a positive effect on pain, posture and the functional state of patients with a fresh vertebral fracture.

The planned study investigates the effect of the orthosis "Spinomed active" in patients aged ≥ 65 years with at least one non-acute osteoporotic vertebral fracture (at least 3 months ago) and chronic back pain.

ELIGIBILITY:
Inclusion Criteria:

* Living independently in the community
* ≥ 1 low-traumatic vertebral fracture ≥ 3 months ago
* Chronic back pain according to the national guideline for low back pain
* Mean back pain intensity NPS ≥ 1 (1-10 scale)
* Hyperkyphosis, kyphosis angle according to Debrunner >40°
* Intact skin or adequate wound coverage in the area of the contact surface of the orthosis

Exclusion Criteria:

* Secondary osteoporosis (as determined by study physician)
* Expected change in overall pain therapy during the study period
* Structurally fixed kyphosis, lack of extension ability of the thoracic spine
* Kyphoplasty, vertebroplasty
* Use of back orthoses during the last 6 months
* Depression
* Dementia, cognitive impairment (Mini Mental Test < 25)
* Fresh neurological deficits; incontinence > grade 1
* Body dimensions that do not allow for adjustment of the back orthosis
* Absence during baseline and follow-up assessments

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes — Higher incidence of osteopenia in female population
Enrollment: 80 (Actual)
Dates: Start 2021-04-07 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2022-01-15 (Actual)

PRIMARY OUTCOMES:
Back pain | At baseline and after 16 weeks (i.e. over 16 weeks)
  Change in back pain (mean intensity over 4 weeks on the "numeric pain scale (NPS) "0-10").

SECONDARY OUTCOMES:
Trunk strength/performance | At baseline and after 16 weeks (i.e. over 16 weeks)
  Changes of maximum dynamic trunk strength (index of trunk extension/flexion/lateral flexion) as determined by a dynamic testing device
Kyphosis angle | At baseline and after 16 weeks (i.e. over 16 weeks)
  Changes of kyphosis angle as determined by angle measurement
Functional capacity | At baseline and after 16 weeks (i.e. over 16 weeks)
  Changes in Chair-Rise-Test
Pulmonary function | At baseline and after 16 weeks (i.e. over 16 weeks)
  Changes in vital capacity as determined by a pulmonary function monitor
Everyday life skills | At baseline and after 16 weeks (i.e. over 16 weeks)
  Changes of everyday life skills as determined by a questionnaire (late-life function and disability instrument)
Balance capacity | At baseline and after 16 weeks (i.e. over 16 weeks)
  Changes in Body Sway as determined by a balance sensor device

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Kemmler, PhD, Study Chair — Institute of Medical Physics, Friedrich-Alexander University of Erlangen-Nürnberg
Locations (1):
- Institute of Medical Physics University of Erlangen-Nurnberg, Erlangen, Germany

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study are available on request from the corresponding researcher (SW)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will become available in March 2022 without time limit.